CLINICAL TRIAL: NCT06652841
Title: Prospective, Multi-center, Single Arm Feasibility Study of the transShield Embolic Protection System
Brief Title: Feasibility Study of the transShield Embolic Protection System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Sponsor closing study due to financial circumstances.
Sponsor: TransAortic Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPL-06-001
Record Dates: First submitted 2024-09-30; First posted 2024-10-22 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Aortic Stenosis
Keywords: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Patients with severe aortic valve stenosis scheduled for TAVR (Experimental): transShield Embolic Protection System
  Interventions: Device: transShield Embolic Protection System

INTERVENTIONS:
Device: transShield Embolic Protection System — Patient undergoing TAVR procedure will receive the transShield EPS with the intent to capture and remove debris dislodged during the interventional procedure.

SUMMARY:
The objective of this study is to evaluate the initial safety and performance of the transShield EPS used for embolic protection during Transcatheter Aortic Valve Replacement (TAVR).

DETAILED DESCRIPTION:
Patients 18 years of age and older, with severe aortic valve stenosis scheduled for a Transcatheter Aortic Valve Replacement (TAVR) procedure will be screened to determine eligibility and interest in the study. Patients who pass pre-screen eligibility criteria and are willing to participate in the study will be asked to sign the study Informed Consent Form before any study-specific tests or procedures are performed or for any study specific evaluations not considered standard of care that need to be performed to assess eligibility. All subjects enrolled in the study will be followed from baseline through post procedure, prior to discharge and conclude with a 30-day followup visit. The investigator will perform the percutaneous TAVR using a commercial TAVR system according to their institution's standard practice. After completion of the procedure, the transShield EPS Filter will be collected and shipped to an independent Core Lab for histopathology assessment of the embolic debris captured in the filter. Post procedure treatment and safety monitoring shall be completed per the investigator's standard guidelines and patients discharged when clinically stable, at the investigator's discretion. Prior to discharge, functional status, physical exam/vital signs, medications, safety assessment and hospital stay information shall be collected. Patients will be asked to return to the investigational site 30 days post procedure for functional status, physical exam/vital signs, medications, and safety assessment. If the patient is not able to return to the investigational site, the visit may be completed via a tele-health visit with the investigator in combination with an in-office visit to the patient's local General Practitioner (GP) or Cardiologist. This visit will conclude the patient's participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥18 years old
2. Patient is scheduled for percutaneous TAVR using a commercial TAVR system
3. Patient meets indications for TAVR per the device IFU
4. The diameter of the artery at the site of the filter placement is ≤ 42 mm
5. Size and condition of the femoral artery iliac arteries are appropriate for the 10F transShield Introducer
6. Patient, or authorized representative, signs a written Informed Consent form to participate in the study, prior to any study mandated procedures
7. Patient is willing and able to complete follow-up requirement

Exclusion Criteria:

1. Patient not undergoing TAVR via the trans-femoral route
2. Carotid artery stenosis > 70% in either carotid artery
3. Severe vascular tortuosity or anatomy that would preclude the safe introduction of the device
4. Aortic valve is a congenital unicuspid valve or is non-calcified
5. Predominant aortic regurgitation >3+
6. A known contraindication or hypersensitivity to all anticoagulation regimens or an inability to undergo anticoagulation for the study procedure
7. History of bleeding diathesis or in whom anticoagulant and/or anti- platelet therapy is contraindicated, patients who will refuse transfusion, or have an active peptic ulcer or upper GI bleeding within the prior 3 months
8. Renal disease requiring chronic dialysis at time of treatment
9. History of stroke or transient ischemic attack (TIA) within prior 6 months
10. Evidence of an acute myocardial infarction (MI) within 30 days prior to study procedure
11. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation, or mechanical heart assistance within prior 30 days
12. Severe left ventricular (LV) dysfunction with LV ejection fraction (LVEF) <20%
13. Severe pulmonary hypertension and right ventricular (RV) dysfunction
14. Echocardiographic evidence of intracardiac mass, thrombus or vegetation
15. Life expectancy <12 months due to non-cardiac co-morbid conditions
16. Evidence of active systemic or local groin infection
17. Significant aortic disease, including abdominal aortic or thoracic aneurysm defined as maximal luminal diameter 5cm or greater; marked tortuosity (hyperacute bend), aortic arch atheroma or severe atheroma (especially with calcification and surface irregularities) of the thoracic aorta, severe "unfolding" and tortuosity of the thoracic aorta
18. Known hypersensitivity or contraindication to aspirin, heparin or bivalirudin, ticlopidine, or clopidogrel, and/or contrast agents, that cannot be managed with premedication
19. Planned other cardiac surgical procedure within 2 weeks prior to or planned cardiac surgical or interventional procedure within 30 days after the TAVR procedure.

    Note: Diagnostic cardiac catheterization is permitted within 10 days prior to the TAVR procedure
20. Known allergy to any device component
21. Known or suspected to be pregnant or lactating
22. Currently enrolled in an investigational drug or device clinical study in which the primary endpoint has not occurred
23. Patient has other medical, social or psychological problem that in the opinion of the investigator precludes them from participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Performance Objective: Technical Success defined as tranShield EPS ability to perform all the following functions without adjudicated device malfunctions: | During procedure
  Ability to successfully deploy the device in the correct anatomical position, in the ascending aorta without interference with TAVR procedure/devices, and ability to retrieve and remove the device intact, including no visual evidence of any filter damage.
Safety Objective: MACCE at 30 Days | 30 day post procedure
  Defined as incidence of Major Adverse Cardiac and Cerebrovascular Events (MACCE) at 30 days according to VARC-3 including: All cause mortality, All stroke (disabling and non-disabling) and TIA, Acute kidney injury (stage 2 or 3), Major vascular and access-related complications, and Life-threatening or disabling bleeding (type 2-4).

SECONDARY OUTCOMES:
Embolic Debris Captured | Procedure
  Volume of debris captured defined as the average number of captured particles great than or equal to 150 µm in diameter, as assessed by independent pathologist.
Incidence of Stroke | Discharge and 30 Day Post-Procedure
  Incidence of stroke according to VARC-3 definitions (subclassified ischemic, hemorrhagic, or undetermined, and as disabling or non-disabling) and TIA
Adverse Events | Up to 30 Days Post-procedure
  Sunmary of all Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Waikato Hospital, Hamilton, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided